CLINICAL TRIAL: NCT01015534
Title: Phase II Randomized Study: Whole Brain Radiotherapy and Concomitant Temozolomide, Compared With Whole Brain Radiotherapy for Brain Metastases Treatment
Brief Title: Whole Brain Radiotherapy With or Without Temozolomide at Daily Fixed-dose for Brain Metastases Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Carlos Gamboa Vignolle, Radiation Oncologist, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 006/004/TEI
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-03

CONDITIONS: Brain Neoplasms
Keywords: Brain metastases; Temozolomide; Whole-brain radiotherapy; Phase II trial
MeSH Terms: conditions — Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole brain irradiation plus Temozolomide (Experimental): Whole brain irradiation at a dose of 30 Gy in 10 daily fractions over 2 weeks, and a fixed dose of oral Temozolomide, 1h before each fraction of whole brain irradiation, 200 mg on Monday, Wednesday, Friday; 300 mg on Tuesday, and Thursday. Without adjuvant cycles of Temozolomide.
  Interventions: Drug: Temozolomide; Radiation: Whole brain irradiation
- Whole brain irradiation (Active Comparator): Whole brain irradiation at a dose of 30 Gy in 10 daily fractions over 2 weeks
  Interventions: Radiation: Whole brain irradiation

INTERVENTIONS:
Drug: Temozolomide
  Other Names: Temodar; or; Temodal
  Arms: Whole brain irradiation plus Temozolomide
Radiation: Whole brain irradiation
  Other Names: Whole brain radiotherapy

SUMMARY:
RATIONALE

* Fractionated radiotherapy uses high-energy photons to kill, or damage tumor cells. High daily dose temozolomide combined with fractionated radiotherapy may make tumor cells more sensible to treatment.

PURPOSE

* This randomized phase II trial, assess in patients with brain metastases from solid tumors, whether the whole brain radiotherapy (WBRT) plus temozolomide is able to improve the results obtained with WBRT.

DETAILED DESCRIPTION:
Primary Outcome Measures

* Objective Response Rates

Secondary Outcome Measures

* Survival Free of Brain Metastases progression
* Overall Survival
* Systemic Side effects

Objectives

Primary

* Compare objective response rates in both arms of treatment

Secondary

* Compare survival free of progression in both arms of treatment
* Compare Overall Survival in both arms of treatment
* Compare side effects

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status (KPS) ≥ 50
* Life expectancy ≥ 12 weeks
* Histologically confirmed non lymphomatous solid tumors at primary site
* Brain metastases diagnosed with cranial MRI/CT.
* Extracranial metastases or primary tumor uncontrolled are allowed
* Hemoglobin ≥ 10 g/dl
* Absolute neutrophil count of > 1500/mm3
* Platelet count of ≥ 100,000/mm3
* Blood urea nitrogen (BUN) ≤ 25 mg/dl,
* Serum creatinin ≤ 1.5 mg/dl
* Serum bilirubins ≤ 1.5 mg/dl,
* Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ twice the upper normal limit

Exclusion Criteria

* Pregnant or breast feeding woman
* History of allergic reaction to iodinated contrast media
* Inability to swallow
* Systemic chemotherapy in previous 3 weeks
* Oral chemotherapy in previous 2 weeks
* Prior surgery, chemotherapy, or radiotherapy for a brain neoplasm
* Meningeal carcinomatosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gamboa-Vignolle, MD, Principal Investigator — Instituto Nacional de Cancerología de México
Locations (1):
- Instituto Nacional de Cancerología de México, México, D.F, Mexico

REFERENCES:
- [Background] Jones SF, Greco FA, Gian VG, Miranda FT, Raefsky EL, Hainsworth JD, Willcutt NT, Beschorner AF, Kennerly G, Burris HA 3rd. A Phase I trial of protracted oral fixed-dose temozolomide. Cancer. 2005 Nov 1;104(9):1985-91. doi: 10.1002/cncr.21408. PMID 16134182
- [Background] Antonadou D, Paraskevaidis M, Sarris G, Coliarakis N, Economou I, Karageorgis P, Throuvalas N. Phase II randomized trial of temozolomide and concurrent radiotherapy in patients with brain metastases. J Clin Oncol. 2002 Sep 1;20(17):3644-50. doi: 10.1200/JCO.2002.04.140. PMID 12202665
- [Background] Verger E, Gil M, Yaya R, Vinolas N, Villa S, Pujol T, Quinto L, Graus F. Temozolomide and concomitant whole brain radiotherapy in patients with brain metastases: a phase II randomized trial. Int J Radiat Oncol Biol Phys. 2005 Jan 1;61(1):185-91. doi: 10.1016/j.ijrobp.2004.04.061. PMID 15629610
- [Derived] Gamboa-Vignolle C, Ferrari-Carballo T, Arrieta O, Mohar A. Whole-brain irradiation with concomitant daily fixed-dose temozolomide for brain metastases treatment: a randomised phase II trial. Radiother Oncol. 2012 Feb;102(2):187-91. doi: 10.1016/j.radonc.2011.12.004. Epub 2012 Jan 16. PMID 22257825

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from patients from Instituto Nacional de Cancerología de México, from January 2006 to September 2008.
Pre-assignment Details: Seventy-two patients were assessed for eligibility. Twelve patients did not meet inclusion criteria. Five patients declined to participate. Fifty-five patients were enrolled.
Groups:
- Whole Brain Irradiation and Temozolomide: Whole brain irradiation, 1 fraction of 3 Gy x 5 days of each week for 2 weeks, Monday to Friday and a fixed dose of oral temozolomide, 1h before each daily fraction of Whole brain irradiation, 200 mg on Monday, Wednesday, Friday; 300 mg on Tuesday, and Thursday. Without extra cycles of Temozolomide.
- Whole Brain Irradiation: Whole brain irradiation, 1 fraction of 3 Gy x 5 days each week for 2 weeks, Monday to Friday.
Period: Overall Study
Arm/Group | Whole Brain Irradiation and Temozolomide | Whole Brain Irradiation
Started | 28 | 27
Completed | 27 | 27
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Whole Brain Irradiation and Temozolomide | Whole Brain Irradiation | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 19 | 44
  >=65 years | 3 | 8 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 49.5 (13.4) | 53.8 (13.7) | 51.7 (13.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  Mexico | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rates. Assessed With Cranial MRI
Description: Objective Response (OR) encompassed the number of participants with Complete Response (CR) and the number of participants with Partial Response (PR). CR is the disappearance of all brain metastases, assessed between two or more cranial MRI. PR is at least a 30% decrease in the sum of the longest diameter of the brain metastases, taking as reference the baseline sum longest diameter, assessed between two or more cranial MRI.
  Objective Response Rate (ORR) is the ratio between the number of participants with objective response and the total number of participants.
Time Frame: 90 days
Population: Data on all enrolled participants were included in an intention-to-treat analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants with OR
Groups:
- Whole Brain Irradiation and Temozolomide: Patients received Whole brain irradiation at a dose of 30 Gy in 10 daily fractions over 2 weeks, and a fixed dose of oral Temozolomide, 1h before each fraction of whole brain irradiation, 200 mg on Monday, Wednesday, Friday; 300 mg on Tuesday, and Thursday. Without adjuvant cycles of Temozolomide.
- Whole Brain Irradiation: Whole brain irradiation,at a dose of 30 Gy in 10 daily fractions over 2 weeks
Arm/Group | Whole Brain Irradiation and Temozolomide | Whole Brain Irradiation
Number analyzed (Participants) | 28 | 27
Percentage of participants with OR | 78.6 [63.4 to 93.8] | 48.1 [29.2 to 66.9]
Statistical Analysis 1: Comparison: Whole Brain Irradiation and Temozolomide vs Whole Brain Irradiation; Test type: Superiority or Other; p = 0.019, Chi-squared — The sample size was calculated with a two-sided test,a type-I error probability of 0.05 and a power of 0.80,Twenty- eight patients in each treatment arm were required to detect a difference in ORR of 0.29; Odds Ratio (OR) = 3.9, 95% CI 2-sided [1.3 to 12.9]

2. Secondary Outcome: Survival Free of Brain Metastases Progression (PFS of BM)
Description: Progression free survival of brain metastases is the survival of participants without progressive brain metastases or without neurological symptoms. The progressive brain metastases (PBM) were evaluated with cranial MRI. The PBM were defined as an increase of at least 20% in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new metastases.
Time Frame: at 90 days
Population: Data on all enrolled participants were included in an intention-to-treat analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Whole Brain Irradiation and Temozolomide: Whole brain irradiation at a dose of 30 Gy in 10 daily fractions over 2 weeks, and a fixed dose of oral Temozolomide, 1h before each fraction of whole brain irradiation, 200 mg on Monday, Wednesday, Friday; 300 mg on Tuesday, and Thursday. Without adjuvant cycles of Temozolomide.
- Whole Brain Irradiation: Whole brain irradiation, at a dose of 30 Gy in 10 daily fractions over 2 weeks
Arm/Group | Whole Brain Irradiation and Temozolomide | Whole Brain Irradiation
Number analyzed (Participants) | 28 | 27
Percentage of Participants | 88.7 [76.7 to 100] | 83.7 [69 to 98.4]
Statistical Analysis 1: Comparison: Whole Brain Irradiation and Temozolomide vs Whole Brain Irradiation; Test type: Superiority or Other; p = .704, Fisher Exact; Odds Ratio (OR) = .688, 95% CI 2-sided [.138 to 3.422]

3. Secondary Outcome: Overall Survival
Description: Overall survival:Time in months measured from treatment initiation until the date of death or the date of last follow-up.
Time Frame: 1 year
Population: Data on all enrolled participants were included in an intention-to-treat analysis.
Measure: Median (95% Confidence Interval); unit: Months of Overall Survival
Arm/Group | Whole Brain Irradiation and Temozolomide | Whole Brain Irradiation
Number analyzed (Participants) | 28 | 27
Months of Overall Survival | 8 [4.9 to 11.1] | 8.1 [5.9 to 10.1]
Statistical Analysis 1: Comparison: Whole Brain Irradiation and Temozolomide vs Whole Brain Irradiation; Test type: Superiority or Other; p = 0.84, Log Rank

4. Secondary Outcome: Number of Grade 3-4 Adverse Events (AE) That Are Definitely or Probably Related to Both Groups of Treatment.
Description: AE, evaluated and graded according to the NCI common terminology criteria (NCI-CTCAE) v3.0
  Grade 3 Severe AE.
  Grade 4 Life-threatening or disabling AE.
Time Frame: 4 months
Population: Participants were assessed with a Complete blood count at the end of the first and second weeks of treatment. A standard biochemical profile was performed at the end of the second week of treatment, at 2 weeks after completion and at 2 months thereafter. Participants also were evaluated clinically with the same periodicity .
Measure: Number; unit: Events
Groups:
- Whole Brain Irradiation and Temozolomide: Whole brain irradiation, Whole brain irradiation at a dose of 30 Gy in 10 daily fractions over 2 weeks,and a fixed dose of oral temozolomide, 1h before each daily fraction of Whole brain irradiation, 200 mg on Monday, Wednesday, Friday; 300 mg on Tuesday, and Thursday. Without extra cycles of Temozolomide.
Arm/Group | Whole Brain Irradiation and Temozolomide | Whole Brain Irradiation
Number analyzed (Participants) | 28 | 27
Events
  Leukopenia | 1 | 0
  Lymphopenia | 11 | 6
  Nausea-Vomiting | 1 | 0
  Neutropenia | 1 | 1
  Platelets | 3 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Patients were assessed as follows: with a Complete blood count at the end of the first and second week of treatment. A standard biochemical profile at the end of the second week of treatment, at 2 weeks after completion and at 2 months thereafter. Also were evaluated clinically with the same periodicity.
Arm/Group | Whole Brain Irradiation and Temozolomide | Whole Brain Irradiation
Serious Adverse Events (participants affected / at risk) | 17/28 | 7/27
Other Adverse Events (participants affected / at risk) | 11/28 | 13/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whole Brain Irradiation and Temozolomide (N=28) | Whole Brain Irradiation (N=27)
Lymphopenia (Blood and lymphatic system disorders) | 11 (11) | 6 (6) — Grade 3 <500 - 200 mm3. Grade 4 <200/mm3
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Grade 3 <2000 - 1000/mm3
Platelets (Blood and lymphatic system disorders) | 3 (3) | 0 (0) — Grade 3 <50,000 - 25,000/mm3. Grade 4 <25,000/mm3
Neutrophils (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Grade 3 <1000 - 500/mm3
Nausea-Vomiting (Hepatobiliary disorders) | 1 (1) | 0 (0) — Grade 3 ≥6 episodes in 24 hrs; IV fluids, indicated ≥24 hrs
OTHER ADVERSE EVENTS (reported when occurring in more than 3.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whole Brain Irradiation and Temozolomide (N=28) | Whole Brain Irradiation (N=27)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 11 (11) — Grade 1 < Low limit of normal (LLN) - 800/mm3. Grade 2 <800 - 500/mm3.
platelets (Blood and lymphatic system disorders) | 3 (3) | 1 (1) — Grade 1 <LLN-75,000/mm3. Grade 2 <75,000-50,000/mm3.
Alanine aminotransferase - Aspartate aminotransferase (Metabolism and nutrition disorders) | 3 (3) | 1 (1) — Alanine aminotransferase Grade 1 > Upper limit of normal (ULN) - 2.5 x ULN Aspartate aminotransferase Grade 1 > ULN - 2.5 x ULN

LIMITATIONS AND CAVEATS:
Our study had methodological limitations, such as the two temozolomide dose levels, which in future clinical trials may be adjusted to a single level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No